CLINICAL TRIAL: NCT05160454
Title: NIRS to Evaluate Haemodynamic Reserve in Paediatric Moyamoya
Acronym: NIRS moyamoya
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16NC24
Record Dates: First submitted 2019-11-08; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Moyamoya
MeSH Terms: conditions — Moyamoya Disease | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: patients and controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Active Comparator): child with moyamoya
  Interventions: Device: near infrared spectroscopy
- control (Active Comparator): unaffected control
  Interventions: Device: near infrared spectroscopy

INTERVENTIONS:
Device: near infrared spectroscopy — evaluate cerebral blood flow with and without breatholding

SUMMARY:
Near infrared spectroscpy is a validated method of evaluating cerebral blood flow. The aim in this pilot study to explore its use in children with moyamoya disease.

DETAILED DESCRIPTION:
Moyamoya disease is a cerebrovascular condition in which there is chronic brain hypoperfusion. As surgery can possibly augment brain blood flow, a method for evalutaing cerebrovascualr reserve would be helpful in selecting patients for intervention.

Near infrared spectroscopy (NIRS) is a validated non-invasive method of evaluating cerebral blood flow. We aim to investigate the feasibility and tolerability of using NIRS haemodynamic reserve in children with moyamoya and controls by evaluating cerebral blood flow in the baseline state and after breath-holding.

Feasibility will be assessed by how many successful studies are carried out. Tolerability will be assessed by asking children some simple questions about their experience.

ELIGIBILITY:
Inclusion Criteria: Patients with moyamoya and unaffected healthy controls -

Exclusion Criteria: age <6

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of NIRS studies that can be completed in moyamoya patients | 2years
  how many studies can be completed

SECONDARY OUTCOMES:
Patient questionnaire to evaluate children's experience of NIRS in moyamoya | 2years
  ask children re their experience

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No